CLINICAL TRIAL: NCT03496389
Title: Does Gabapentin Reduce Quadriceps Muscle Weakness After Anterior Cruciate Ligament Reconstruction? A Randomised Controlled Trial
Brief Title: Does Gabapentin Reduce Quadriceps Muscle Weakness After Anterior Cruciate Ligament Reconstruction?
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Ng Jonathan Patrick, Principle investigator, Hospital Authority, Hong Kong
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Gabapentin ACLR
Record Dates: First submitted 2018-03-29; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Muscle Weakness; Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Muscle Weakness; Anterior Cruciate Ligament Injuries | interventions — Gabapentin; Tramadol; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Gabapentin + panadol (Experimental)
  Interventions: Drug: Gabapentin; Drug: Panadol
- Tramadol + panadol (Active Comparator)
  Interventions: Drug: Tramadol; Drug: Panadol

INTERVENTIONS:
Drug: Gabapentin — Gabapentin 300mg daily
  Arms: Gabapentin + panadol
Drug: Tramadol — Tramadol 50mg QID
  Arms: Tramadol + panadol
Drug: Panadol — Panadol 500mg QID

SUMMARY:
Anterior cruciate ligament (ACL) injury is a common sport injury in both professional and recreational athletes. Furthermore, persistent quadriceps weakness and wasting are frequently observed after anterior cruciate ligament reconstruction (ACLR). Several studies have demonstrated that muscular rehabilitation to normal strength is difficult, protracted, and often not achieved due to the inability to fully activate the quadriceps voluntarily. Pain and disuse are often blamed for the inhibition of muscle activation following joint injury. However, arthrogenic muscle inhibition (AMI) is often overlooked and not addressed. Thus, the magnitude of strength restoration of the quadriceps is frequently restricted despite solid rehabilitation protocols. As AMI is a reflex inhibition of musculature involving the neurotransmitter γ-aminobutyrate (GABA), Gabapentin may have a potential role in modulating AMI, therefore limiting muscle weakness after ACLR.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50
2. Unilateral isolated ACL tear for primary ACLR confirmed clinically and radiologically
3. No concomitant ligamentous, meniscal or chondral injuries.

Exclusion Criteria:

1. Concomitant multiple ligament injuries including posterior cruciate ligament, medial collateral ligament ligament, or lateral collateral ligament
2. Concomitant meniscal injuries
3. Concomitant chondral injuries
4. preoperative radiographic signs of arthritis
5. Revision ACL surgery
6. Contralateral knee with
7. Medical co-morbidities including Diabetes Mellitus, chronic renal failure
8. Documented hypersensitivity to Gabapentin
9. History of epilepsy
10. History of depression
11. Non-compliance to rehabilitation protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in from baseline quadriceps muscle strength | at postoperative 4, 6, 9, 12 months
  Will be measured using Biodex isodex dynamometer to measure peak torque of knee extension

SECONDARY OUTCOMES:
Anterior-posterior knee stability | at postoperative 4, 6, 9, 12 months
  Measured by Lachman test
Anterior-posterior knee stability | at postoperative 4, 6, 9, 12 months
  Measured by anterior drawer test
Anterior-posterior knee stability | at postoperative 4, 6, 9, 12 months
  Measured by KT- 1000 knee arthrometer
Rotational laxity | at postoperative 4, 6, 9, 12 months
  Measured using the pivot shift test according to the IKDC score
Functional outcome | at postoperative 4, 6, 9, 12 months
  Measured using single leg hop test
Functional outcome | at postoperative 4, 6, 9, 12 months
  Measured using Lysholm knee scoring system

IPD SHARING:
Plan to Share IPD: Undecided